CLINICAL TRIAL: NCT00337831
Title: Clinical Study on Optimised Removal of Protein-bound Uremic Toxins With Convective Dialysis Treatment.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Gambro Corporate Research, Sweden (Other)
Responsible Party: Natalie Meert, University Hospital Ghent
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2006/127
Record Dates: First submitted 2006-06-15; First posted 2006-06-16 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Renal Failure
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Performance of predilution hemofiltration, predilution hemodiafiltration or postdilution hemodiafiltration — Performance of predilution hemofiltration, predilution hemodiafiltration or postdilution hemodiafiltration is followed.

SUMMARY:
Patients will be treated with hemodiafiltration (HDF) in postdilution mode, as a control therapy, during 9 weeks. During week 5 the 1st intervention treatment, predilution hemofiltration (HF) or predilution HDF, will be performed as a midweek session. After 4 additional weeks of control therapy the other intervention treatment will be performed. Samples will be taken during week 4, 5 and 9: from inlet blood flow (0, 30, 60, 120 and 240 min), from outlet blood flow and dialysate outflow (30, 60, 120 and 240 min).

ELIGIBILITY:
Inclusion Criteria:

* stable on hemodialysis >= 6 months
* of which presently on high-flux HD >= 1 month
* 18 years < age < 85 years
* blood flow rate >= 300ml/min

Exclusion Criteria:

* expected survival < 1 year
* expected transplant within < 1 year
* infectious diseases
* pregnancy
* chronic inflammation condition
* treated with single needle dialysis
* presently treated with hemodiafiltration or low-flux hemodiafiltration
* expected intradialytic body weight gain >= 4kg

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-05; Primary Completion 2007-02 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
To evaluate what is more effective for convective removal of protein-bound solutes - predilution or postdilution of blood? | Samples taken at week 4, 5 and 9. Bloodsamples taken at 0, 30, 60, 120 and 240 min. Dialysate taken at 30, 60, 120 and 240 min.
To check which respective roles diffusion and convection play in the removal of protein-bound uremic toxins? | Samples taken at week 4, 5 and 9. Bloodsamples taken at 0, 30, 60, 120 and 240 min. Dialysate taken at 30, 60, 120 and 240 min.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Vanholder, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be